CLINICAL TRIAL: NCT03333135
Title: The Pulmonary Consequences of Participating in the UTMB and Hong Kong 100 Ultramarathons and Impact of Phased Electromagnetic Field Therapy (PEMF)
Brief Title: Ultramarathons and Impact of Phased Electromagnetic Field Therapy (PEMF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Johnson, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-003843
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Ultramarathons; Electromagnetic field therapy; Endurance; Exercise; Environmental conditions
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study team and participants will not know if they have received the PEMF therapy or the sham
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HK100 Pulsed Electromagnetic Field (Experimental): 20 athletes (ideally a mix of elite and amateur level athletes and veteran (40-65y) and young (20-39y). Athletes will be recruited at the 2018 and 2019 Hong Kong 100 races. In addition, these athletes will use the pulsed electromagnetic field (PEMF) for the two weeks prior to the race.
  Interventions: Procedure: Pulsed Electromagnetic Field therapy (PEMF)
- HK100 Pulsed Electromagnetic Field Sham (Sham Comparator): 20 athletes (ideally a mix of elite and amateur level athletes and veteran (40-65y) and young (20-39y). Athletes will be recruited at the 2018 and 2019 Hong Kong 100 races. In addition, these athletes will use a PEMF device that doesn't produce electromagnetic fields (sham) for the two weeks prior to the race.
  Interventions: Procedure: Pulsed Electromagnetic Field Sham therapy
- UTMB Pulsed Electromagnetic Field (Experimental): 20 athletes (ideally a mix of elite and amateur level athletes and veteran (40-65y) and young (20-39y). Athletes will be recruited at the 2018 and 2019 Ultra Trail du Mont Blanc (UTMB) races. In addition, these athletes will use the pulsed electromagnetic field (PEMF) for the two weeks prior to the race.
  Interventions: Procedure: Pulsed Electromagnetic Field therapy (PEMF)
- UTMB Pulsed Electromagnetic Field Sham (Sham Comparator): 20 athletes (ideally a mix of elite and amateur level athletes and veteran (40-65y) and young (20-39y). Athletes will be recruited at the 2018 and 2019 Ultra Trail du Mont Blanc (UTMB) races. In addition, these athletes will use a PEMF device that doesn't produce electromagnetic fields (sham) for the two weeks prior to the race.
  Interventions: Procedure: Pulsed Electromagnetic Field Sham therapy

INTERVENTIONS:
Procedure: Pulsed Electromagnetic Field therapy (PEMF) — PEMF Therapy based on Biological Electromagnetic (BEM) microbial wave technology provides micro-magnetic emissions to the center of the palm (Laogong acupoint). While participating in the study, the subjects will undertake 2 sessions of therapy every day (1 session in the morning and evening). Each session will last for 16-min (8-min for left and 8-min for right hand).
  Other Names: Bioboosti
  Arms: HK100 Pulsed Electromagnetic Field; UTMB Pulsed Electromagnetic Field
Procedure: Pulsed Electromagnetic Field Sham therapy — PEMF therapy will be administered however it will not produce micro-magnetic emissions. The therapy will be used on the center of the palm (Laogong acupoint) of each hand. While participating in the study, the subjects will undertake 2 sessions of therapy every day (1 session in the morning and evening). Each session will last for 16-min (8-min for left and 8-min for right hand).
  Other Names: Bioboosti Sham
  Arms: HK100 Pulsed Electromagnetic Field Sham; UTMB Pulsed Electromagnetic Field Sham

SUMMARY:
This research is being done to better understand the pulmonary consequences of completing an ultra marathon at altitude and a sea level city.

DETAILED DESCRIPTION:
Subjects will be asked to undertake three (3) sets of assessments at prescribed time intervals: Baseline (at 72-24h prior to each event), immediately post (within 2h of race completion) and during recovery (within 24-48h of race completion). Each assessment will consist of 1)lung function tests; 2) a saliva and blood sample; 3) a lung and cardiac ultrasound. Subjects will be recruited from a range of age groups and fitness levels, before being divided into a sham or therapy group. Groups will use Pulsed Electromagnetic Field (PEMF) therapy or related sham before the event and during recovery.

ELIGIBILITY:
Inclusion Criteria:

Healthy endurance trained individuals participating in the Ultra Trail du Mont Blanc (UTMB) and/or Hong Kong 100 ultramarathons

Exclusion Criteria:

> 65 years age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in right ventricle end diastolic area (EDA) | baseline, within 2 hours of race completion, 24-48 hours post race
  Cardiac ultrasound (Philips CX50) will be performed to determine left and right ventricular morphology and function. Ultrasound will be performed in accordance with the recommendations of the American Society of Echocardiography guidelines (ASE). Imaging of the ventricles and the diameter during relaxation (diastole) will be captured and evaluated. Normal value for right ventricle EDA indexed to body surface area ranges between 5-12.6 cm^2/m^2 for males and 4.5-11.5 cm^2/m^2 for females .
Change in tricuspid annular plane systolic excursion (TAPSE) | baseline, within 2 hours of race completion, 24-48 hours post race
  Another ultrasound metric that will be evaluated is tricuspid annular plane systolic excursion (TAPSE) which is used a parameter of global RV function which describes apex-to-base shortening. Normal value for TAPSE is above 16 mm.
Change in ratio between early mitral inflow velocity and mitral annular early diastolic velocity (E/e') | baseline, within 2 hours of race completion, 24-48 hours post race
  Another ultrasound metric that will be evaluated is early mitral inflow velocity and mitral annular early diastolic velocity (E/e') which is used to evaluate the diastolic or relaxation function of the left ventricle. Normal value for E/e' is <6.
Change in the ratio of peak velocity flow in early diastole (the E wave) to peak velocity flow in late diastole caused by atrial contraction (the A wave) | baseline, within 2 hours of race completion, 24-48 hours post race
  Another ultrasound metric that will be evaluated is he ratio of peak velocity flow in early diastole (the E wave) to peak velocity flow in late diastole caused by atrial contraction (the A wave) (E/A) which is used to evaluate the diastolic filling of the left ventricle. Normal value for E/A is between 0.8 and 2.
Change in lung fluid assessed through ultrasound incidence of comet tails | baseline, within 2 hours of race completion, 24-48 hours post race
  Ultrasound will be used to image 28 "windows" covering the 2nd through the 5th intercostal/rib space on the right and left sides of the chest. The number of comet tails observed over these 28 locations will be documented and the change in this number over the course of the study will be evaluated.
Change in lung fluid assessed through diffusion capacity of the lungs for carbon monoxide and nitric oxide | baseline, within 2 hours of race completion, 24-48 hours post race
  Subjects will take a maximal breath of a test gas mixture, hold that inhalation for 4 seconds and then exhale and the exhaled gas will be analyze to determine the change in gas concentrations between what was inhaled and exhaled. Comparison will be made between the change over time in this ability of gas to move from the lungs to the blood stream.

SECONDARY OUTCOMES:
Change in exhaled nitric oxide | baseline, within 2 hours of race completion, 24-48 hours post race
  The amount of nitric oxide in ones exhaled air will be measured by a handheld device. Levels under 25 parts per billion are normal, more than 35 parts per billion would be a sign of airway inflammation.
Change in hemoglobin | baseline, within 2 hours of race completion, 24-48 hours post race
  A blood sample will be taken and analyzed to determine the amount of red blood cells and and hemoglobin in the blood. For males normal range for hemoglobin is 13.5-17.5 grams per deciliter and for females normal range for hemoglobin is 12.0-15.5 grams per deciliter. Low values means anemia is present and higher levels is a normal response to altitude.
Change in hematocrit | baseline, within 2 hours of race completion, 24-48 hours post race
  A blood sample will be taken and analyzed to determine the amount of red blood cells and and hemoglobin in the blood. For males normal range for hematocrit is 38.8-50% and for females normal range for hematocrit is 34.9-44.5% Low values means anemia is present and higher levels is a normal response to altitude.
Change in cardiac troponin I | baseline, within 2 hours of race completion, 24-48 hours post race
  To determine if signs of cardiac damage, as its presence in the blood is a potential sign of damage to the heart muscle
Change in B-type natriuretic peptide | baseline, within 2 hours of race completion, 24-48 hours post race
  To determine if signs of cardiac damage, as its presence in the blood is a potential sign of damage to the heart muscle
Change in cortisol | baseline, within 2 hours of race completion, 24-48 hours post race
  Saliva levels of cortisol will be measured as a metric of stress. Cortisol levels increase when you body is under stress.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials